CLINICAL TRIAL: NCT00306761
Title: Effects of Dynamic Wheelchair Seating on Spasticity and Functional Mobility in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Michael E. Hahn, Assistant Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSU_Thrasher
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dynamic Wheelchair Seating System

SUMMARY:
Cerebral palsy (CP) is a non-degenerative neuromuscular disease that can exist at or occur as a result of birth. Because of damage to one or more parts of the brain that control movement, an affected child cannot control his or her muscles normally. Prevalence of CP is similar worldwide, with pronounced severity in underdeveloped countries due to poor health and financial conditions.

Research should be conducted to find methods of medical treatment to allow affected children to maintain or regain musculoskeletal functionality. Many children affected with CP spend much of their days restricted to a rigid wheelchair; limiting muscular and cognitive development, making it difficult to interact with their environment. The gap to be addressed by this study is to determine if a wheelchair that is based on the dynamics of human anatomy can allow enhanced function, while being adaptive to individual growth and development. At present, there is very little dynamic capability available in commercial wheelchairs to allow this mobility.

A dynamic wheelchair system was recently designed and a small sample of able-bodied children has been tested in the chair. It is hypothesized that significant increases in functional mobility will be achieved in children with CP from the use of this novel wheelchair design.

DETAILED DESCRIPTION:
Specifically, it is expected that range of motion and functional mobility in the hip, knee, and ankle joints will increase, involuntary spasticity in the musculature of the mid and lower body will be reduced, and independent daily function will be enhanced in children with CP. The success of these conditions will greatly influence the child's interaction with the surrounding environment, maintaining neuromuscular function and providing enhanced mobility for coordinated development through childhood.

This research will bring great benefits for children with CP, however children with other neuromuscular conditions should also benefit from the findings of this initial study. Specifically, the direct health benefits will include increased joint range of motion, reduction of spasticity, enhanced cognitive development and muscle coordination. The concept of this novel wheelchair design could be applied domestically within one year of project completion. If funded, this initial study will lead to a subsequent project of two years, which would focus on the feasibility of broadening the target population to include children in under-represented areas within the United States and in developing countries.

Twenty children (4-12 years) with CP will be recruited for this study from the surrounding community and greater Rocky Mountain region. The study volunteers will be randomly assigned to either an experimental group (using new dynamic seating system), or a control group (using standard, state of the art non-dynamic chair systems). Consent will be obtained from each child and their parents/guardians. The study will consist of a pre-chair laboratory session, a supervised chair adaptation period (including a mid-way laboratory session) and a follow-up laboratory session. The pre-chair, mid-way and follow up laboratory sessions will consist of a series of cognitive/communicative, fine motor, and functional skill tests. Evaluation of these tests will be conducted by physical, occupational, and speech therapists. The wheelchair effect will be tested for significant improvement in joint range of motion, muscle spasticity and tone, and independent functionality.

ELIGIBILITY:
Inclusion Criteria:

* Spastic Cerebral Palsy
* Requires Wheelchair for mobility

Exclusion Criteria:

* Unable to respond to clinical evaluation commands

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Joint range of motion
Muscle spasticity
Functional Capacity Assessments

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Hahn, PhD, Principal Investigator — Montana State University
Locations (1):
- Epicenter Therapy Services, Bozeman, Montana, United States